CLINICAL TRIAL: NCT03619915
Title: Correlation Between Spirometry and Functional Independence in Adult Post-ICU Patients
Status: Completed | Type: Observational
Sponsor: Universidade Estadual do Oeste do Paraná (Other)
Responsible Party: Principal Investigator, Pericles Almeida Delfino Duarte, MD, PhD, Clinical Professor of Department of Medicine, Western Parana State University Hospital, Universidade Estadual do Oeste do Paraná
Other Study IDs: 436.770-1
Record Dates: First submitted 2018-07-20; First posted 2018-08-08 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Intensive Care (ICU) Myopathy; Functional Independence
MeSH Terms: conditions — Muscular Diseases | interventions — Spirometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Greater dependence
  Interventions: Diagnostic Test: Spirometry; Other: Functional Independence Measure
- Less dependence
  Interventions: Diagnostic Test: Spirometry; Other: Functional Independence Measure
- Independent
  Interventions: Diagnostic Test: Spirometry; Other: Functional Independence Measure

INTERVENTIONS:
Diagnostic Test: Spirometry — The test will follow the norms of the American Thoracic Society and reference values relative to the Brazilian population. The tests will be performed by physical therapists using the One Flow FVC® portable spirometer (Clement Clarke, England) and met the criteria for acceptance and reproduction of manoeuvres
Other: Functional Independence Measure — Will be used to evaluate the functional independence of patients containing eighteen items encompassing six dimensions. Each item can receive scores of one to seven, where one corresponds to total dependency and seven to full independence. Each dimension is analysed by the sum of the items that compose it and the total score is given by the sum of each dimension, being able to vary from 18: complete dependence; 19 to 60: greater dependence (assistance of up to 50% of tasks); 61 to 103: less dependency (assistance of up to 25% of tasks); and 104 to 126: independent.

SUMMARY:
Several complications and comorbidities are frequently found in patients admitted to an Intensive Care Unit (ICU), including acquired ICU muscle weakness and physical and cognitive limitations. These issues lead to impaired quality of life and post-discharge functional independence. Thus, it is important to evaluate these factors in order to verify the effects of long-term hospitalization. Objective: To relate functional independence to the degree of pulmonary involvement in adult patients three months after discharge from the ICU. Methods: This will be a retrospective study with data collected from January 2012 to December 2013, that will include patients who underwent spirometry and answered the Functional Independence Measure Questionnaire. Patients will be divided into groups according to the classification of functional independence and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients who discharged alive evaluated three months after discharge from the ICU
* Patients that underwent spirometry and answer the Functional Independence Measure Questionnaire.

Exclusion Criteria:

* Patients unable to perform spirometry
* Patients unable to respond to the Functional Independence Measure questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from patients admitted to the ICU from January 2012 to December 2013.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Spirometry | Three months after ICU discharge
  The spirometry will follow the norms of the American Thoracic Society and reference values relative to the Brazilian population. The tests will be performed by physical therapists using the One Flow FVC® portable spirometer (Clement Clarke, England) and met the criteria for acceptance and reproduction of manoeuvres.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | Three months after ICU discharge
  FIM will be use to evaluate the functional independence of patients containing eighteen items encompassing six dimensions. Each item can receive scores of one to seven, where one corresponds to total dependency and seven to full independence. Each dimension is analysed by the sum of the items that compose it and the total FIM score is given by the sum of each dimension, being able to vary from 18: complete dependence; 19 to 60: greater dependence (assistance of up to 50% of tasks); 61 to 103: less dependency (assistance of up to 25% of tasks); and 104 to 126: independent.